CLINICAL TRIAL: NCT00003780
Title: An Open Label Randomized Trial Comparing the Safety and Efficacy of Systemic Chemotherapy (Gemcitabine) to Immunotherapy (CYTOIMPLANT - Intra Tumor Implants of Allogeneic Peripheral Blood Mononuclear Cells Sensitized Against Patient Alloantigens by Mixed Lymphocyte Culture) as First Line Therapy for Patients With Unresectable Locally Advanced, and Metastatic Pancreatic Cancer
Brief Title: Chemotherapy Compared to Biological Therapy in Treating Patients With Cancer of the Pancreas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meyer Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066912; MEYER-AIT-PAN-201
Record Dates: First submitted 1999-11-01; First posted 2004-09-14 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-05

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

INTERVENTIONS:
Biological: tumor infiltrating lymphocyte therapy
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. It is not yet known whether chemotherapy is more effective than biological therapy in treating patients with cancer of the pancreas.

PURPOSE: Randomized phase II trial to compare the effectiveness of gemcitabine with biological therapy in treating patients who have cancer of the pancreas that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of CYTOIMPLANT (intratumor implants of allogeneic peripheral blood mononuclear cells sensitized against patient alloantigens by mixed lymphocyte culture) vs gemcitabine in patients with unresectable, locally advanced or metastatic pancreatic cancer. II. Compare the overall survival, progression free survival, objective tumor response, time to treatment failure, and quality of life of these patients. III. Compare the safety and toxicities of CYTOIMPLANT vs gemcitabine in these patients.

OUTLINE: This is a randomized, open label, multicenter study. Patients are randomly assigned (2:1 ratio in favor of CYTOIMPLANT arm) to one of two treatment arms. Arm I: Patients receive gemcitabine IV weekly for 7 weeks, followed by 1 week of rest. In subsequent courses, patients then receive gemcitabine IV weekly for 3 weeks followed by a week of rest. Courses are repeated every 4 weeks in the absence of disease progression or unacceptable toxicity. Arm II: Patients undergo leukapheresis to collect lymphocytes. Patient lymphocytes are mixed with donor lymphocytes at the sponsor labs. The mixture is implanted into the tumor using endoscopic ultrasound guided fine needle injection. This process may be repeated in the fifth month using different donor's lymphocytes. Follow up assessments may include physical exams, lab tests, CT scans, and quality of life assessments at 4 weeks and at 3, 5, 7, 9, and 12 months from the date of randomization. Patients are then contacted every 3 months to assess status.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage II, III, or IV pancreatic cancer that is unresectable No symptomatic third space fluid collection (e.g., ascites, pleural effusion)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 3 months Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hematocrit at least 33% Hemoglobin at least 10.5 g/dL Hepatic: Bilirubin no greater than 3.0 mg/dL SGOT or SGPT no greater than 3 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No history of myocardial infarction within past 3 months No congestive heart failure Other: HIV negative No other prior malignancy except basal cell skin cancer No persistent fever greater than 102 degrees F (39 degrees C) unless caused by the pancreatic cancer Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy (e.g., interferons, interleukins) Chemotherapy: No prior chemotherapy Endocrine therapy: No concurrent systemic steroids Radiotherapy: No prior radiotherapy Surgery: At least 30 days since prior surgery Decompressive surgery and endoscopic stenting (including expandable wire stents) allowed to relieve symptoms of disease Other: At least 30 days since prior investigational therapy Palliative care to relieve symptoms of disease allowed, including pain management and celiac block by endoscopic ultrasonography or percutaneously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 1998-12

CONTACTS AND LOCATIONS:
Overall Officials: Michael F. O'Neill, Study Chair — Meyer Pharmaceuticals
Locations (1):
- Meyer Pharmaceuticals, LLC, Irvine, California, United States